CLINICAL TRIAL: NCT01663441
Title: Multicenter, Randomized Phase Ⅲa Study of Genetically Modified Recombinant Human Interleukin-11 to Prevent Chemotherapy-induced Thrombocytopenia in Cancer Patients Receiving Chemotherapy.
Brief Title: A Phase Ⅲa Study of Genetically Modified Recombinant Human Interleukin-11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NL201-Ⅲ-2012
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2017-07

CONDITIONS: Chemotherapy-induced Thrombocytopenia
Keywords: Chemotherapy; Thrombocytopenia; Interleukin-11; Platelet
MeSH Terms: conditions — Thrombocytopenia | interventions — oprelvekin; Interleukin-11; Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Experimental): Patients in this treatment group will receive NL201(5μg/kg) in the first Chemotherapy cycle.Then，in the second Chemotherapy cycle，receive NL201(7.5μg/kg).
  Only for Dose-finding in Phase Ⅲa.
  Interventions: Drug: NL201
- A2 (Experimental): Patients in this treatment group will receive NL201(7.5μg/kg) in the first Chemotherapy cycle.Then，in the second Chemotherapy cycle，receive NL201(5μg/kg).
  Only for Dose-finding in Phase Ⅲa.
  Interventions: Drug: NL201
- A (Active Comparator): Patients in this treatment group will receive NL201（optimal dosing dose）in the first Chemotherapy cycle.Then，in the second Chemotherapy cycle，receive rhIL-11(25μg/kg).
  Only in Phase Ⅲb.
  Interventions: Drug: NL201; Drug: rhIL-11
- B (Active Comparator): Patients in this treatment group will receive rhIL-11(25μg/kg) in the first Chemotherapy cycle.Then，in the second Chemotherapy cycle，receive NL201（optimal dosing dose）.
  Only in Phase Ⅲb.
  Interventions: Drug: NL201; Drug: rhIL-11

INTERVENTIONS:
Drug: NL201 — mIL-11:5μg/kg，subcutaneous administration once daily for 10 days,beginning 24 h after chemotherapy；
  Other Names: mIL-11
  Arms: A1; A2
Drug: NL201 — mIL-11:7.5μg/kg，subcutaneous administration once daily for 10 days,beginning 24 h after chemotherapy；
  Other Names: mIL-11
  Arms: A1; A2
Drug: NL201 — The optimal dosing dose NL201，subcutaneous administration once daily for 10 days,beginning 24 h after chemotherapy.
  Other Names: mIL-11
  Arms: A; B
Drug: rhIL-11 — rhIL-11(25μg/kg)，subcutaneous administration once daily for 10 days,beginning 24 h after chemotherapy.
  Other Names: Recombinant Human Interleukin-11 for Injection
  Arms: A; B

SUMMARY:
This phases Ⅲ trials is divided into two stages,Ⅲa and Ⅲb.The aim of Ⅲa is to evaluate the optimal dosing dose of genetically modified recombinant human IL-11 (mIL-11) in a multicenter randomized self-control trial involving 60 cancer patients undergoing chemotherapy.The aim of Ⅲb is to evaluate the efficacy and safety of genetically modified recombinant human IL-11 (mIL-11), using rhIL-11 as an active control, in a multicenter randomized trial involving 240 cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
The investigators recently developed a mutant form of rhIL-11 with improved stability. In in vitro experimental systems, mIL-11 was shown to endure chemical and proteolytic stresses more effectively, while retaining the biological activity of the original rhIL-11. The improved stability of mIL-11 was also demonstrated in the comparative pharmacokinetic study of subcutaneously delivered mIL-11 and rhIL-11 in the rodent and primate models. Based on its improved pharmacokinetic and pharmacodynamic features. In Phase II study shows that mIL-11 is well tolerated and has thrombopoietic activity equivalent to one third of the clinical dose of rhIL-11, indicating the potential of mIL-11 for use in the treatment of CIT. This study is a phase III, single-blinded, randomized,multicenter,cross-over study designed to evaluate optimal dosing dose and efficacy and safety of mIL-11 on CIT patients receiving suitable chemotherapeutic regimen for treating cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological verification of malignancy at the time of initial diagnosis；
* Patients (age,18-75 years) receiving chemotherapy, who had experienced platelet counts below 75×10^9/L；
* patients were required to have adequate bone marrow,hepatic, and renal functions at the time of study entry；
* ECOG ≤2；
* patients to have normal laboratory findings:while white blood count >3.0×10^9/L,platelet count ≥100×10^9/L, and AST and/or ALT lesser than 2.5 times the upper limit of the normal value；
* The estimated life expectancy of the patient was more than 3 months.

Exclusion Criteria:；

* patients who received total body irradiation；
* patients with childbearing potential；
* patients who were breast-feeding or pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Recovery time of platelet counts from below 100x10^9/L raise to more than 100 x10^9/L. | During 21 days of chemotherapy cycles

SECONDARY OUTCOMES:
Nadir platelet counts | During 21 days of chemotherapy cycles
Platelet counts at day 21 after the initiation of chemotherapy. | Day 21 after the initiation of chemotherapy.
Average platelet counts | During 21 days of chemotherapy cycles
Incidence of thrombocytopenia | During 21 days of chemotherapy cycles

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- See also: Related Info — http://www.northland-bio.com/